CLINICAL TRIAL: NCT03891797
Title: PTSD Treatment for Incarcerated Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0630; A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Processing Therapy (Experimental): 12 sessions of group-based Cognitive Processing Therapy administered 1x/week for 90 minutes each session.
  Interventions: Other: Cognitive Processing Therapy
- Control (No Intervention): No treatment/treatment as usual. Participants will complete questionnaires at three time points with no intervention.

INTERVENTIONS:
Other: Cognitive Processing Therapy — Group-based psychotherapy.
  Other Names: CPT
  Arms: Cognitive Processing Therapy

SUMMARY:
There is a particular need for more effective treatments for post-traumatic stress disorder (PTSD) within the incarcerated population. The prevalence of trauma history and PTSD are markedly higher in jail and prison populations than in the general population, with estimates of current PTSD prevalence among prison inmates exceeding 20%, as opposed to 3-6% in the general population. Cognitive Processing Therapy (CPT) is a potentially promising PTSD treatment for the prison setting.

The primary objectives of this project include:

1. Establish the feasibility of group CPT delivery in male and female prisons with PTSD by examining participant retention in the 12-week course;
2. Obtain preliminary efficacy estimates for reducing PTSD symptom severity, as well as secondary symptoms associated with trauma, including depression, hopelessness, self-blame, and negative self-related thoughts.

DETAILED DESCRIPTION:
PTSD is associated with an increased risk for crime-related behaviors, such as violence and substance abuse. There is virtually no research examining the efficacy of empirically-supported therapies for PTSD in incarcerated individuals. Despite the patent need for more effective treatment strategies, there is scant translational research on PTSD in the criminal offender population, and no randomized controlled studies that have tested the efficacy of empirically-supported PTSD treatments in the prison setting. The treatment programs offered to prison inmates (across the United States, but particularly in Wisconsin) target specific, overt criminal behaviors (e.g., alcohol/drug use, violence, sexual offenses), rather than underlying psychopathology. Our program of research could usher a new paradigm of offender rehabilitation, by addressing the traumatic experiences and consequent psychopathology that predispose individuals to certain forms of maladaptive and criminal behavior.

Cognitive Processing Therapy (CPT) is a potentially promising PTSD treatment for the prison setting, primarily due to its cost- and time-effectiveness in the manualized group format. Individual (one-on-one) therapies such as Prolonged Exposure and Eye Movement Desensitization and Reprocessing are less likely to gain widespread implementation in prison systems, where therapist access is a major limitation. In addition, CPT is applicable to a wide range of individuals, such as those with minimal formal education, low intelligence (IQs), or comorbid psychiatric disorders. In studies of non-incarcerated individuals, CPT has been found to be more effective than wait-list control and equivalent to Prolonged Exposure. The majority of non-incarcerated individuals undergoing CPT for PTSD exhibit a clinically significant reduction in symptoms, with over 40% achieving a loss of the diagnosis. However, the generalizability of these findings to the offender population has not yet been determined. This research study will determine whether CPT is indeed an effective and feasible treatment for PTSD in inmates, or whether different treatment strategies need to be developed.

Hypotheses:

Regarding Aim 1, it is predicted that feasibility will be established by obtaining ≥80% participant retention for the CPT course. Additional metrics of feasibility will assess eligibility; participation; compliance; adherence; competence; and safety.

Regarding Aim 2, it is predicted that PTSD symptom reduction will be greater among CPT participants than waitlist control participants. Furthermore, it is predicted that reductions in depression, hopelessness, self-blame, and negative self-related thoughts will also be greater in the CPT group.

This study will screen approximately 100 participants for eligibility over 2 years. Over the two-year study, two 12-week sessions of CPT will be run in each of the two prisons (one housing male offenders and one housing female offenders).

A total of 64 inmates (32 male and 32 female) will participate in group randomization. In order to generate a sufficient pool of eligible subjects who meet inclusion criteria for the study, approximately 200 inmates per year will be interviewed and screened (100 male and 100 female per year) during the two-year study period (400 total screened for eligibility; 64 total enrolled in the study).

Research Design and Procedures:

Potential participants will be contacted by calling them over the phone system within the prison. Potential participants arrive to a private testing room and are asked if they would like to learn about the study and potentially participate. If so, the consent process will begin.

Eligible participants will first complete the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (SCID-5) to ascertain current PTSD symptomology and diagnosis. This assessment will take approximately 1-2 hours. Participants may have recently completed the SCID-5 as part of a separate study (2014-1106 "Neuropsychological screening and testing for University of Wisconsin (UW)-Department of Corrections (DOC) collaborative research project"). Participants who have completed the SCID-5 as part of study 2014-1106 less than two months from the time of enrollment for this study will not complete the SCID-5 again, the SCID-5 information obtained from study the PI's database will be used.

Participants will then be assigned to CPT or a control group. The CPT group will engage in 12, 90-minute treatment sessions (18 hours total). CPT group-members are asked to complete weekly homework (approximately 12 hours total). Approximately 8 participants will be included in each CPT session. Participants with PTSD will be randomized to the CPT group or control group. Participants will be notified via institutional mail when they are starting CPT, or if they have been randomized to the control group. The control group will be asked to complete the same pre-, mid- and post-treatment questionnaires as the CPT group, but they will not engage in the study intervention. Participants in the control group will be able to continue any ongoing treatment/interventions they are engaged in within the institution. All participants will be asked what treatment groups they are currently enrolled in during the initial screening to examine the possibility of attentional bias within the CPT group (i.e., more frequent interaction leading to treatment outcomes).

The control group will be asked to complete three sessions in total (pre-, mid-, and post-testing), and will complete these assessments on the same timeline as the CPT group (described above).

Initial assessment and study consent will be conducted by trained graduate students and/or advanced undergraduates with extensive experience working on our prison project. All treatment groups will be conducted by an advanced graduate student in the clinical psychology program, with supervision provided by a licensed clinical psychologist.

Treatment notes will be completed after each group session to document the content covered in the group and to track the attendance of group members. Group members will not receive individual psychotherapy notes, and no information from this study will be added to participants' medical record.

To ensure that the randomization process results in CPT and control group that are balanced on key variables that might affect treatment response, participants will be assigned to groups through stratified randomization, in which randomization occurs within specific strata of different potential moderating variables and assures equal assignment to each group across these variables. Participants will be stratified/randomized based on PTSD scores. IQ and age will be included as covariates in all analyses.

Treatment:

The CPT group will include up to 8 members and will meet weekly for 12 sessions in total. Participants will be referred to by their preferred first names. The CPT protocol will follow the published manual. Session 1 begins with education about PTSD, an overview of treatment, and an assignment to write an impact statement about the personal meaning of the traumatic event. After reading and discussing the meaning of the traumatic event in Session 2, group members are introduced to the identification of and relationship among events, thoughts, and emotions. At the end of Session 3, group members are given the assignment of recording events, thoughts, and emotions throughout the week to establish the relationships between thoughts and emotions within their own lives. During Session 4, cognitive therapy begins with Socratic questions regarding self-blame and other distortions regarding the event. In Sessions 5-6, the focus of the therapy shifts to teaching clients to challenge and change their beliefs about the meaning of the event and the implications of the trauma for their lives. Group members are first taught to challenge a single thought by asking themselves a series of questions. They are then taught to identify problematic patterns of cognition that have come to represent a style of responding. From that point, beginning with Session 7, group members use worksheets that incorporate the earlier activities as well as the development of alternative, more balanced self-statements. In Sessions 7-12, group members are asked to focus on one of the five core themes of CPT each week (safety, trust, power-control, esteem, or intimacy) and correct any overgeneralized beliefs related to that theme. In Session 11, group members are asked to rewrite their impact statements to reflect their current beliefs, and these revised statements are then used in Session 12 to evaluate gains made in treatment and areas in which they wish to continue working.

The therapist for the CPT group has master's level training in clinical psychology. She will be trained through 16 hours of initial individual training plus five additional hours over the course of the treatments (21 hours total). This level of training emulates the personnel and training resources that would realistically be available in the correctional setting (i.e., to make the results of this research program generalizable and scalable to correctional institutions). Training will be provided by a licensed clinical psychologist with experience in student supervision and clinical research and with particular expertise in CPT. This level of therapist training is believed to be sufficient for this project, as a previous study showed group CPT to be effective for reducing PTSD symptoms in a resource-poor country where the therapists had minimal secondary education and the patients had extremely limited literacy.

ELIGIBILITY:
Inclusion Criteria:

* DSM 5 criteria for current PTSD diagnosis
* IQ greater than 70
* Reading level of 5th grade or higher
* No history of psychosis or dementia
* Stable medication use (same medication for at least one month) if using medication
* No scheduled transfer or release for at least 12 weeks (the duration of the intervention).

Exclusion Criteria:

* Other vulnerable populations within the prison setting will not be eligible for participation, such as:

  * pregnant women
  * individuals who have English as a second language
  * those with visual or hearing impairments
  * individuals appearing to lack the capacity to provide informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
PTSD-Checklist-5 (PCL-5) | 4 months
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Participants rate on a 0 ("not at all") - 4 ("Extremely") scale how bothered they have been by PTSD symptoms in the last month. Total scores range from 0-80.
Eligibility | 3 months
  Percentage of inmates who meet the full set of inclusion criteria.
Participation | 4 months
  Percentage of eligible inmates agreeing to participate in randomization into one of the two groups.
Retention | 12 weeks
  Percentage of inmates attending all 12 sessions.
Compliance | 4 months
  Compliance will be measured in three ways: Percentage of retained inmates performing intervention activities during session (e.g., attending to and contributing to the discussion); the percentage of inmates completing the homework assignment each week; and the percentage of inmates fully completing the pre-, mid-, and post-intervention assessment batteries. All three measures of compliance will be reported individually. An overall metric of compliance will be calculated by averaging the three individual measures.
Adherence | 12 weeks
  Adherence will by measured by the presence or absence of five session elements (scores 0-5) by the clinical supervisors, as in previous CPT studies.
Competence | 12 weeks
  Ratings of the quality of session elements (scores 1-7; 1="not satisfactory", 4="satisfactory", 7="excellent") by the clinical supervisors, as in previous CPT studies
Safety-Suicidal ideation item on the Beck Depression Inventory-II (BDI-II) | 4 months
  The BDI-II is a 21-item self-report questionnaire assessing symptoms of depression in the last 2-weeks. Each item is on a 0-3 scale, with higher scores indicative of greater symptom severity. Scores range from 0-63.

SECONDARY OUTCOMES:
Posttraumatic Cognition Inventory (PCTI) | 4 months
  The PCTI is a 33-item self-report questionnaire that assesses on a scale from 1(totally disagree) to 7 (totally agree) individuals agree with trauma-related maladaptive beliefs (e.g., "I am a weak person"). Scores range from 33-231.
Beck Hopelessness Scale (BHS) | 4 months
  The BHS is a 20-item self-report questionnaire assessing symptoms of hopelessness. Each item is a "true" or "false statement. Scores range from 0-20 depending on the number of items endorsed in the hopelessness direction.
Beck Depression Inventory (BDI-II) | 4 months
  The BDI-II is a 21-item self-report questionnaire assessing symptoms of depression in the last 2-weeks. Each item is on a 0-3 scale, with higher scores indicative of greater symptom severity. Scores range from 0-63.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koenigs, PhD, Principal Investigator — UW-Madison
Locations (1):
- Fox Lake Correctional Institute, Fox Lake, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Informed consent gives permission to share de-identified participant data (all primary and secondary outcome measures) with other UW-Madison researchers. Other data sharing is not currently approved.

REFERENCES:
- [Background] Goff A, Rose E, Rose S, Purves D. Does PTSD occur in sentenced prison populations? A systematic literature review. Crim Behav Ment Health. 2007;17(3):152-62. doi: 10.1002/cbm.653. PMID 17595672
- [Background] Egeressy A, Butler T, Hunter M. 'Traumatisers or traumatised': Trauma experiences and personality characteristics of Australian prisoners. Int J Prison Health. 2009;5(4):212-22. doi: 10.1080/17449200903343209. PMID 25757522
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Kilpatrick DG, Resnick HS, Milanak ME, Miller MW, Keyes KM, Friedman MJ. National estimates of exposure to traumatic events and PTSD prevalence using DSM-IV and DSM-5 criteria. J Trauma Stress. 2013 Oct;26(5):537-47. doi: 10.1002/jts.21848. PMID 24151000
- [Background] Elbogen EB, Johnson SC, Wagner HR, Sullivan C, Taft CT, Beckham JC. Violent behaviour and post-traumatic stress disorder in US Iraq and Afghanistan veterans. Br J Psychiatry. 2014;204(5):368-75. doi: 10.1192/bjp.bp.113.134627. Epub 2014 Feb 27. PMID 24578444
- [Background] Campbell CA, Albert I, Jarrett M, Byrne M, Roberts A, Phillip P, Huddy V, Valmaggia L. Treating Multiple Incident Post-Traumatic Stress Disorder (PTSD) in an Inner City London Prison: The Need for an Evidence Base. Behav Cogn Psychother. 2016 Jan;44(1):112-7. doi: 10.1017/S135246581500003X. Epub 2015 Feb 20. PMID 25697197
- [Background] Heckman CJ, Cropsey KL, Olds-Davis T. Posttraumatic stress disorder treatment in correctional settings: A brief review of the empirical literature and suggestions for future research. Psychotherapy (Chic). 2007 Mar;44(1):46-53. doi: 10.1037/0033-3204.44.1.46. PMID 22122167
- [Background] Resick, P.A., C.M. Monson, and K.M. Chard, Cognitive Processing Therapy for PTSD: A Comprehensive Manual. 2016: Guilford Press.